CLINICAL TRIAL: NCT07320469
Title: Efficacy of Inspiratory Muscle Trainer on Respiratory Functions Exercise Capacity and Pain Intensity in Adults With Obesity and Mechanical Low Back Pain. A Randomized Clinical Trial.
Brief Title: Efficacy of Inspiratory Muscle Trainers on Patients With Obesity and LowBack Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Maali Mohammed Alqahtani, Lecturer, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: IRB-PGS-2025-03-0528
Record Dates: First submitted 2025-11-16; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Obesity; Low Back Pain
Keywords: obesity; low back pain; obesity and low back pain; inspiratory muscle trainers; respiratory function; exercise capacity; functional disability; pain intensity; body compisition
MeSH Terms: conditions — Obesity; Low Back Pain; Respiratory Aspiration; Pain

STUDY DESIGN:
Intervention Model Description: The study design will be a parallel-group, double-blind, randomised controlled trial.After referral from the orthopedic or neurology clinic to the Respiratory Care (RC) Department, participants will undergo screening for low back pain to include only those diagnosed with mechanical low back pain. Following this, the assessor will record each participant's demographic data, including gender, age, BMI, blood pressure (BP), heart rate (HR), duration of pain, and pain severity using the Numerical Pain Rating Scale (NPRS). A Bioelectrical Impedance Analysis (BIA) device will be used to measure fat-free mass, fat percentage, and body cell mass before and after the training intervention (Schoeller, 2000). Baseline measurements will be taken prior to the intervention and again after six weeks by a blinded assessor.
Who Masked: Participant, Outcomes Assessor
Masking Description: Each participant will be stratified and assigned either to a control or experimental group based on age, pain score and BMI.
  Blinding & Randomization will be performed by computer-generated numbers from www.randomizer.org. A random number generator will make a serial number for each participant. Both participants and the assessor will be blinded. Participants will be randomized into the experimental group; they will practice an aerobic exercise and resistance training program in addition to IMT with resistance set at 40% of each participant's maximum inspiratory pressure, while all participants of the control group will practice aerobic exercise and resistance training in addition to IMT with no resistance (Ponde et al., 2021 & Medicine, 2014).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group : IMT with 40%Of MIP +walking +resisancee training (Experimental): Experimental Group: Twenty-four participants will practice aerobic exercise (30 minutes of walking at 40-60% of HRmax) and resistance training in addition to IMT (starting resistance level of 40%) three times a week for six weeks.
  Home program: All participants of both groups will also perform different exercises, including aerobic, resistive, and IMT training two times per week at home. The participants from both groups will receive detailed instructions to guide them in performing home sessions. Follow up with them through WhatsApp and Zoom, and call them every other day to check their performance and encourage them. Participants will also have logbooks for documentation and to count the adherence and compliance.
  Interventions: Device: Inspiratory muscle trainer
- Control group: IMT with 0% of MIP +walking +resistance training (Placebo Comparator): Twenty-four participants will practice aerobic exercise (30 minutes of walking at 40-60% of HRmax) and resistance training in addition to IMT (starting resistance level of 0%) three times a week for six weeks.
  Home program: All participants of both groups will also perform different exercises, including aerobic, resistive, and IMT training two times per week at home. The participants from both groups will receive detailed instructions to guide them in performing home sessions. Follow up with them through WhatsApp and Zoom, and call them every other day to check their performance and encourage them. Participants will also have logbooks for documentation and to count the adherence and compliance.
  Interventions: Device: Inspiratory muscle trainer

INTERVENTIONS:
Device: Inspiratory muscle trainer — Inspiratory muscle trainer: The POWER breath device has a variable resistance, which can be adjusted by a calibrated spring. The initial resistance training level will be adjusted at 0% resistance for the control group and 40% of MIP for the experimental group. The participants will be instructed to use the device twice daily (two times per day, in the hospital under supervision, 30 breaths in each session) for three days a week for 6 weeks, with periods of rest, especially if the patient feels dizzy or fatigued.

SUMMARY:
Background: Obesity and mechanical low back pain (MLBP) are two major health problems negatively affecting the human body. Many studies have shown that obesity and MLBP are associated with negative effects on the respiratory system. There are many interventions to treat obesity and MLBP, such as aerobic exercise and diet programs. Moreover, the Inspiratory Muscle Trainer (IMT) significantly improved inspiratory muscle strength in patients with obesity. This study aims to investigate whether adding IMT to aerobic exercise will improve respiratory function, exercise capacity, and pain intensity in patients with obesity and MLBP. Materials and Methods: A total of forty-eight obese patients with MLBP will be equally and randomly assigned to the experimental group and control group. The experimental group will have training on IMT for 6 weeks, three days per week (two sessions daily, thirty breaths per session) using POWERbreathe IMT, starting at 40% of maximal inspiratory pressure with increasing training load at the third week, in addition to having aerobic exercise three times a week for 30 minutes and total body resistance. The control group will have the same training as the experimental group, except for IMT; they will have zero resistance. Main outcome measures: pulmonary function tests and maximal inspiratory pressures to assess respiratory function; VO2 to assess exercise capacity; pain intensity; and Oswestry Disability Index to determine functional disability. All the measurements will be done before and after the intervention in both groups. Paired and independent t-tests will be used to compare within- and between-group differences. A repeated-measures design will be used to determine significant differences before, during, and after the intervention within each group.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effects of inspiratory muscle trainers on respiratory function, exercise capacity, pain intensity, and functional disability in patients with obesity and MLBP. If a significant improvement is found, IMT could be added to the guidelines for exercise prescriptions for obese patients with MLBP. Therefore, this study might provide evidence-based findings to guide clinical decision-making and empower clinicians and healthcare organizations to incorporate IMT into exercise prescription guidelines for obese patients with MLBP. By integrating IMT into guidelines, this study might enhance rehabilitation strategies for obese patients with MLBP.

Hypothesis

* Null Hypothesis: the addition of IMT to aerobic exercise does not result in significant differences in respiratory functions, exercise capacity, pain intensity, and functional disability in patients with obesity and mechanical low back pain.
* Alternative Hypothesis: the addition of IMT to aerobic exercise results in significant differences in respiratory functions, exercise capacity, pain intensity, and functional disability in patients with obesity and mechanical low back pain.

Objectives of the study:

1. To assess the effects of PowerBreathIMT on pulmonary function tests and maximum inspiratory pressure in patients with obesity and mechanical low back pain.
2. To assess the effects of PowerBreathIMT on exercise capacity, pain intensity and functional disability in patients with obesity and mechanical low back pain.

Expected Results The addition of IMT to aerobic exercise results in significant differences in respiratory functions, exercise capacity, pain intensity, and functional disability in patients with obesity and mechanical low back pain.

Material and methods:

o Study setting: The current study will be conducted at King Fahad Hospital of the University, Al Khobar, Saudi Arabia. All participants will be recruited from the orthopedic and neurological clinics after confirming their diagnosis (they suffer from mechanical low back pain & exclude the existence of other causes for back pain). All measurements will be done at the Pulmonary Function Test Lab in the previous week of our intervention and in the next week after the end of our intervention. Participants will practice the supervised sessions at the hospital three times per week for six weeks. During supervised sessions, all participants will follow a dietary regime and perform aerobic exercise and resistance training in addition to IMT training.

NB: Home program: All participants of both groups will also perform aerobic exercise and IMT training two sessions per week at home. The participants from both groups will receive detailed instructions to guide them in performing home sessions. A follow-up with them will be through WhatsApp and Zoom, and I will call them every other day to check their performance. The participants will also have logbooks to document aerobic exercise, resistance training, and IMT training at home and to document the adherence and completeness of the training program.

NB: Diet Program: All participants of both groups will follow an individualized diet program.

* Sample Size Calculation: Sample size was calculated by using data from a previous study that assessed the significant difference between two independent means (intervention and control groups) with a primary outcome measure of Vital Capacity from a Pulmonary Function Test (mean 1 = 4.28 and mean 2 = 4.07, sigma= 0.2) . The parameters used for the calculation included an alpha level of 0.05 and a power of 0.90. This link was used, which is a valid and reliable tool for calculating sample size when comparing two means. The sample size was 20 participants in each group to find out a significant difference with sufficient power. So, the total sample size will be 40. However, to account for a 20% attrition rate and dropouts, the sample size will be adjusted. The adjusted sample size will be calculated as a total of 48 participants, resulting in approximately 24 participants in each group.

  • Ethical considerations: Ethical approval was obtained from the institutional review board of the Dean of Scientific Research at Imam Abdulrahman bin Faisal University. Moreover, approval from the Saudi Food and Drug Administration was obtained. Each patient will sign a consent form to authorize participation. They will be informed that their information and data will be confidential, and the collected data will be published in the future. The participants will be informed that participation is voluntary, and they can withdraw at any time without consequences.
* Recruitment and study population: Participants who meet the inclusion criteria will be recruited from orthopedic and neurologic clinics in the outpatient department of King Fahad Hospital of the University to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Aged between 20 and 50 years
* Obese and experiencing mechanical low back pain (MLBP)
* A body mass index (BMI) between 30 and 40 kg/m²
* low back pain for more than 12 weeks, with pain localized to the lumbar region - A pain score greater than 3 but less than 7 on the Numeric Pain Rating Scale (NPRS).
* Low back pain will be screened using the Mechanical and Inflammatory Low Back Pain (MIL) Index.
* Stable and controlled medical conditions

Exclusion Criteria:

* Medically unstable
* Severe spinal pathology, e.g., infection, tumor, arthritis, inflammation, spine deformity, advanced neurologic diseases, head or spinal surgeries, rheumatic diseases, and respiratory muscle paralysis
* Acute inflammation of the musculoskeletal system
* Pregnancy
* Unable to follow instructions, e.g., those with learning difficulties

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Function Test | 6 weeks
  a. Pulmonary Function Tests: are essential for assessing lung function and are highly valid and reliable. Spirometry will be used to assess pulmonary function following standard maneuvers.
Maximal Inspiratory Pressure | 6 weeks
  b. Maximum Inspiratory Pressure (MIP) is a reliable and valid measure of inspiratory muscle strength, influenced by factors such as age, sex, height, and weight. It demonstrates good test-retest reliability and strong concurrent validity when compared with reference tests in COPD patients. It will be measured by cmH₂O.

SECONDARY OUTCOMES:
Maximal O2 uptake (VO2 max) | 6 weeks
  a. Maximal O₂ uptake (VO₂ max) is the gold standard for assessing cardiovascular fitness and aerobic capacity, showing excellent validity and reliability. VO₂ max reflects the efficiency of the cardiovascular and respiratory systems in oxygen delivery and utilization. It is measured by ml/kg/min.
Pain intensity | 6 weeks
  Pain intensity will be assessed using the 11-point Numerical Pain Rating Scale (NPRS), ranging from 0 ("no pain") to 10 ("worst imaginable pain"). The NPRS shows excellent reliability and strong validity.
Body composition | 6 weeks
  Body composition will be measured using a bioelectrical impedance analyzer (BIA), which estimates body composition by measuring the body's impedance to a small electrical current. By using personal data, the device provides valid and reliable measurements across populations. The measurement will be by Body Mass Index, which is expressed as KG/M². BIA assessments will be conducted before and after training to compare changes in body composition.
Oswestry Disability Index (Arabic Version) | 6 weeks
  The questionnaire will be administered to both groups before and after the intervention. It is a valid and reliable tool that assesses the impact of back pain on daily activities. It includes 10 sections covering various life aspects, including pain intensity. Scores are interpreted as follows: 0-20% = minimal disability, 21-40% = moderate disability, 41-60% = severe disability, and 81-100% = exaggerated symptoms and severe impairment, requiring urgent intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Maali M Alqahtani, Master, Principal Investigator — Imam Andulrahman BinFaisal University; Alsayed M Shanab, PhD, Study Director — Imam Abdulrahman BinFaisal University